CLINICAL TRIAL: NCT02701413
Title: Vaginal Electrical Stimulation for Postpartum Neuromuscular Recovery
Acronym: VESPR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Evergreen Invitational (Unknown)
Responsible Party: Principal Investigator, Christina Lewicky-Gaupp, Assistant Professor, Department of Obstetrics & Gynecology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STU00201026
Record Dates: First submitted 2016-02-10; First posted 2016-03-08 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Obstetric Anal Sphincter Injury; Vaginal Electrical Stimulation
Keywords: Apex M; Postpartum; Pelvic Floor rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ApexM Device (Experimental): The ApexM Device (InControl Medical) is a cylindrical inflatable instrument with electrodes on the dorsal and ventral sides. It is a battery operated, non-implanted device which will be inserted into the vagina and will stimulate the pelvic floor muscles. This device has been shown to be safe and effective for clinical use. Stimulation will alternate between 13 and 50Hz. The initial intensity will be set by the clinician at the patient's initial visit and will be increased in a standard fashion over the duration of the trial.
  Interventions: Device: ApexM (Stimulation) Device
- Sham Device (Sham Comparator): The ApexM Device will be identical in every way but the electrical stimulation will be disabled. The device will still turn on and inflate to fit the contours of the vagina.
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: ApexM (Stimulation) Device — Vaginal electrical stimulation will be administered via the Apex M Device. During each session, the patient will be supine, place conductive gel on the device, insert the device into the vagina, and inflate it to comfort. Subsequently, the device will be turned on and set to previously determined setting. Stimulation session will last 10 minutes and occur 6 times per week for a total of 12 weeks.
  Arms: ApexM Device
Device: Sham Device — A sham Apex M device without electrical stimulation will be used. During each session, the patient will be supine, place conductive gel on the device, insert the device into the vagina, and inflate it to comfort. Subsequently, the device will be turned on and set to previously determined setting. Each session will last 10 minutes and occur 6 times per week for a total of 12 weeks.
  Arms: Sham Device

SUMMARY:
For too many women, childbirth results in devastating consequences: involuntary loss of feces or urine (fecal or urinary incontinence). In fact, up to 50 percent of women with severe tears during childbirth may develop these problems. These new mothers avoid leaving home in order to stay close to a toilet, wear protective pads every day, and avoid activities they previously enjoyed such as exercise and sexual intercourse. It is not surprising that many of these women suffer from postpartum depression, and bonding with their newborns is compromised.

Fecal and urinary incontinence occur due to injuries to the pelvic nerves and muscles during childbirth. Many researchers have focused on what can be done to prevent these injuries; however, few have investigated how to help the countless women who have already suffered from these injuries to the nerves and muscles. In other fields such as orthopedics and neurology, research shows that electrical stimulation can provoke nerve regeneration after injury. Applying this technology to women who have recently suffered from nerve injury during childbirth could have profound and life-changing effects. Investigators hypothesize that electrical stimulation immediately postpartum will markedly help pelvic nerves regenerate, minimizing rates of fecal and urinary incontinence for this vulnerable population of new mothers.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous (First delivery)
* Women who sustain Obstetric Anal Sphincter Injury (OASIS) during first vaginal delivery
* Between age of 18 - 50 years
* English speaking and reading

Exclusion Criteria:

* Implanted electrical device or cardiac arrhythmia
* Neurological disorder
* Inflammatory bowel disease
* Chronic Steroid Use
* Wound breakdown and infection
* Anticipated geographic relocation

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-02-26; Primary Completion 2019-12 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Lewicky-Gaupp, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Medical Group's Integrated Pelvic Health Program, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rockwood TH, Church JM, Fleshman JW, Kane RL, Mavrantonis C, Thorson AG, Wexner SD, Bliss D, Lowry AC. Patient and surgeon ranking of the severity of symptoms associated with fecal incontinence: the fecal incontinence severity index. Dis Colon Rectum. 1999 Dec;42(12):1525-32. doi: 10.1007/BF02236199. PMID 10613469
- [Derived] Brown O, Heliker BD, Geynisman-Tan J, Tavathia M, Mueller MG, Collins S, Kenton K, Lewicky-Gaupp C. Vaginal Electrical Stimulation for Postpartum Neuromuscular Recovery: A Randomized Clinical Trial. Female Pelvic Med Reconstr Surg. 2021 Nov 1;27(11):659-666. doi: 10.1097/SPV.0000000000001037. PMID 34608032

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ApexM Device | Sham Device
Started | 33 | 33
Completed | 26 | 22
Not Completed | 7 | 11
Not completed — Withdrawal by Subject | 7 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ApexM Device | Sham Device | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (4) | 34 (4) | 33 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 9 | 0 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 21 | 32
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Anal Incontinence
Description: The FISI is a validated instrument for assessing fecal incontinence symptom severity. The questionnaire contains 4 questions that assess the frequency of incontinence of solid stool, liquid stool, mucus and gas. FISI total scores range from 0-61 points and higher scores on the scale indicate greater severity of anal incontinence symptoms (worse symptoms). The following are ranges of the scores for each subscale, similarly higher scores on the scale indicate greater severity of subtype of anal incontinence (worse symptoms) Gas subscale- 0-12 points Mucus subscale: 0- 12 points Liquid stool subscale: 0-19 points Solid stool subscale: 0-18 points There are units for the scores on the scale. The Total FISI score is derived from the sum of all the scores on the subscales.
Time Frame: 13 weeks postpartum
Population: Between February 2016 and September 2018, 48 women completed 13-week follow up.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 26 | 22
Scores on a scale | 12 [0 to 23] | 4 [0 to 10]
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Urinary Incontinence
Description: Stress Urinary Incontinence will be compared between the electrical stimulation and sham group by comparing the proportion of women who answer "yes" to the question that corresponds to the presence of stress urinary incontinence (question 17) on the validated questionnaire (Urinary Distress Inventory - 6 (UDI-6).
Time Frame: 1 week postpartum and 13 weeks postpartum
Population: Between February 2016 and September 2018, 30 women completed the UDI-6 at two time points (1 week & 13 week postpartum).
Measure: Count of Participants; unit: Participants
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 13 | 17
Participants
  1 week Post Partum | 8 | 8
  13 Week Postpartum | 5 | 9

3. Secondary Outcome: Number of Participants With Levator Ani Muscle Defects on Either Side of the Pelvis
Description: Endovaginal ultrasound will be used to determine the relationship between levator ani muscle defects between the electrical stimulation and sham group.
  We defined levator ani defect as the separation (avulsion) of any of the levator muscles from one of their primary attachment sites on ultrasound.
  For levator ani defects, the presence or absence of levator ani avulsion (separation from the pubic bone) will be noted on each side. Number of patients with and without these avulsions defects will be compared between the two groups.
Time Frame: 13 weeks postpartum
Population: Between February 2016 and September 2018, 48 women completed 13-week follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 26 | 22
Participants | 8 | 7

4. Secondary Outcome: Number of Patients With Anal Sphincter Muscle Defects
Description: For anal sphincter muscle defects, the number of patients with anal sphincter muscles (out of 360 degrees) will be reported. The proportion of patients with anal sphincter defects in each group will be compared between the two groups.
Time Frame: 13 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 26 | 22
Participants | 12 | 10

5. Secondary Outcome: Maximum Squeeze Anal Pressure
Description: Anal manometry will be used to obtain the maximum squeeze pressures and this will be compared between the electrical stimulation and sham group. Anorectal manometry was performed using a microtipped transducer anorectal manometry system with Laborie software and a 4-channel Gaeltec catheter (Laborie Medical Technologies Co., Williston, VT, and Unisensor, Inc, Hampton, NH). Maximum squeeze pressures at 1, 2, 3, 4, and 5cm proximal to the anal verge were recorded in the semi recumbent position. Maximum squeeze pressure was defined as the highest pressure recorded above the baseline (zero) at any level of the anal canal during maximum squeeze effort by the patient
Time Frame: 13 weeks postpartum
Population: Between February 2016 and September 2018, 48 women completed 13-week follow up.
Measure: Mean (Standard Deviation); unit: mm/Hg
Arm/Group | ApexM Device | Sham Device
Number analyzed (Participants) | 26 | 22
mm/Hg | 108.4 (36.2) | 113.3 (17.7)
Statistical Analysis 1: Comparison: ApexM Device vs Sham Device; Test type: Other; p = 0.88, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 12 weeks of study participation (Baseline= 1 week postpartum and the end point was 13 weeks postpartum) starting from February 2016 and ending in September 2018.
Arm/Group | ApexM Device | Sham Device
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 2/26 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ApexM Device (N=26) | Sham Device (N=22)
UTI (Infections and infestations) | 1 (1) | 0 (0) — Urinary Tract Infection, unknown if related to device use
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Pain with device use

LIMITATIONS AND CAVEATS:
Approximately 27% of the enrolled participants dropped out before study completion. Therefore we had incomplete outcome data for these individuals which introduces attrition bias. Second, the study also was not powered to the secondary outcomes and results from our secondary analyses should be interpreted with this consideration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT02701413/Prot_SAP_000.pdf